CLINICAL TRIAL: NCT06132763
Title: Addressing Root Causes of Under-hydration in School: A Stakeholder Collaborative Pilot Study
Brief Title: Healthy Hydration Pilot in Elementary Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20023592
Record Dates: First submitted 2023-10-31; First posted 2023-11-15 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Hydration; Dental Caries; Body Mass Index
Keywords: Hydration; Water bottle; Sugary Beverages
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydration Intervention (Experimental): Students and staff at the intervention school will receive a school-based hydration intervention that includes a student-developed marketing campaign and incentivizes water bottles in school.
  Interventions: Behavioral: Hydration Intervention
- Control (Placebo Comparator): Students and staff at the control school will participate in assessments only.
  Interventions: Other: Control - Assessments Only

INTERVENTIONS:
Behavioral: Hydration Intervention — Teacher & student ambassadors: serve as hydration role models, identify "Hydration Heroes", monitor filter lights on hydration stations, & update the water meter visual.
  Kick-off event: event to kick off the hydration intervention to include water bottles distribution with a station to personalize, experiential activities, and information about the intervention.
  Social marketing: student-developed marketing campaign "Make water your superpower" will be placed in high-traffic areas of the school. Hydration Headquarters will be located in the lunchroom displaying a water meter illustrating bottle refills from the school's hydration stations.
  Behavioral reinforcement: on random days, students drinking water and/or with a water bottle will receive small incentives.
  Education and outreach: Hydration Tip Sheets, hydration signage in classrooms, and hydration trivia on hydration stations. Teachers will deliver 1 hydration lesson per month that align with Standards of Learning.
  Arms: Hydration Intervention
Other: Control - Assessments Only — Assessments only
  Arms: Control

SUMMARY:
This study will pilot a school-based stakeholder-informed hydration intervention and examine its feasibility and preliminary efficacy.

DETAILED DESCRIPTION:
Adequate water intake plays an important role in maintaining children's overall health, cognitive performance, fine motor skills and visual attention. It also plays a role in the maintenance of healthy weight. Many children do not consume sufficient water, especially in school. There is also potential that by providing enhanced access to water, there will be corresponding decreases in sugary beverage intake. Sugary beverages have been implicated as major contributors of excessive sugar and calorie intake in children, leading to multiple health concerns, such as type 2 diabetes, overweight and obesity, and dental caries. Schools are an optimal environment to increase children's water intake. Healthy hydration is a priority for Richmond Public School (RPS), as they recently adopted a new hydration policy into their school wellness policy, with hydration stations installed in all RPS schools. The purpose of this study is to determine the feasibility of a school-based hydration intervention. This study will pilot a school-based stakeholder-informed hydration intervention and examine its feasibility and preliminary efficacy.

ELIGIBILITY:
Inclusion:

* Lunchroom observations: All students (K-5th) who eat lunch in the cafeteria on assessment days are eligible for lunchroom observations (observing what beverages are selected and presence of water bottles)
* BMI and dental caries assessments: 1) student is in the 3rd grade; 2) English or Spanish speaking.
* Student surveys: Students in 4th-5th grade are eligible to complete surveys assessing beverage intake and perceptions of hydration practices in their district.
* Staff surveys: All staff in the target schools will be eligible to complete the School Environment Survey.

Exclusion:

* Lunchroom observations: None.
* BMI and dental caries assessments: Students are ineligible if they: 1) are non-English or non-Spanish speaking; 2) have a medical condition that precludes drinking water or that can put them at risk for failure to thrive or poor weight gain, 2) are unable to complete assessments due to developmental delays, 3) plan to move from the school district during the study period.
* Student surveys: Students in 4th-5th grade who are unable to complete surveys due to developmental delays will be ineligible.
* Staff surveys: None.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Bean, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two matched schools were randomly selected and assigned to either Intervention or Control group in Fall 2023. Thus, the students and personnel at each school were randomly assigned to the same group as the school they attended/worked at.
  Schools participated in study activities throughout the 2023-2024 school year. A subset of the student population, third graders, were recruited to participate in biomedical assessments (anthropometrics and dental exams).
Units Other Than Participants: School
Groups:
- Hydration Intervention - Students: Students at the intervention school will receive a school-based hydration intervention that includes a student-developed marketing campaign and incentivizes water bottles in school.
  Hydration Intervention: Teacher & student ambassadors: serve as hydration role models, identify "Hydration Heroes", monitor filter lights on hydration stations, & update the water meter visual.
  Kick-off event: event to kick off the hydration intervention to include water bottles distribution with a station to personalize, experiential activities, and information about the intervention.
  Social marketing: student-developed marketing campaign "Make water your superpower" will be placed in high-traffic areas of the school. Hydration Headquarters will be located in the lunchroom displaying a water meter illustrating bottle refills from the school's hydration stations.
  Behavioral reinforcement: on random days, students drinking water and/or with a water bottle will receive small incentives.
  Education and outreach: Hydration Tip Sheets, hydration signage in classrooms, and hydration trivia on hydration stations. Students will receive 1 hydration lesson per month that align with Standards of Learning.
- Hydration Intervention - Personnel: Staff at the intervention school will receive a school-based hydration intervention that includes a student-developed marketing campaign and incentivizes water bottles in school.
  Hydration Intervention: Teacher & student ambassadors: serve as hydration role models, identify "Hydration Heroes", monitor filter lights on hydration stations, & update the water meter visual.
  Kick-off event: event to kick off the hydration intervention to include water bottles distribution with a station to personalize, experiential activities, and information about the intervention.
  Social marketing: student-developed marketing campaign "Make water your superpower" will be placed in high-traffic areas of the school. Hydration Headquarters will be located in the lunchroom displaying a water meter illustrating bottle refills from the school's hydration stations.
  Behavioral reinforcement: on random days, students drinking water and/or with a water bottle will receive small incentives.
  Education and outreach: Hydration Tip Sheets, hydration signage in classrooms, and hydration trivia on hydration stations. Teachers will deliver 1 hydration lesson per month that align with Standards of Learning.
- Control - Students: Students at the control school will participate in assessments only.
  Control - Assessments Only: Assessments only
- Control - Personnel: Staff at the control school will participate in assessments only.
  Control - Assessments Only: Assessments only
Period: Overall Study
Arm/Group | Hydration Intervention - Students | Hydration Intervention - Personnel | Control - Students | Control - Personnel
Started | 278; 1 School | 25; 1 School | 232; 1 School | 28; 1 School
Completed | 278; 1 School (This number reflects the total number of students enrolled and participated in cafeteria observations and school personnel who provided consent to complete personnel surveys. Because the majority of data are de-identified and observation only, we are unable to report if enrollment changed at post. Two students did not participate in post biomedical assessments, but were still enrolled as students and may have participated in observational assessments.) | 25; 1 School | 232; 1 School (This number reflects the total number of students enrolled and participated in cafeteria observations and school personnel who provided consent to complete personnel surveys. Because the majority of data are de-identified and observation only, we are unable to report if enrollment changed at post.) | 28; 1 School
Not Completed | 0; 0 School | 0; 0 School | 0; 0 School | 0; 0 School

BASELINE CHARACTERISTICS:
Population: Number of students enrolled, number of staff that completed a baseline survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydration Intervention - Students | Hydration Intervention - Personnel | Control - Students | Control - Personnel | Total
Number analyzed (Participants) | 278 | 25 | 232 | 28 | 563
Age, Categorical [Count of Participants; unit: Participants] — Population: Age data were pre-specified to not be collected for this study for personnel
  Participants
    number analyzed (Participants) | 278 | 0 | 232 | 0 | 510
    <=18 years | 278 |  | 232 |  | 510
    Between 18 and 65 years | 0 |  | 0 |  | 0
    >=65 years | 0 |  | 0 |  | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 149 | 0 | 119 | 0 | 268
  Sex: Female | 129 | 0 | 113 | 0 | 242
  Sex: Unknown/Not Reported | 0 | 25 | 0 | 28 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black, not of Hispanic origin | 154 | 0 | 101 | 0 | 255
  Race/Ethnicity: White, not of Hispanic origin | 70 | 0 | 87 | 0 | 157
  Race/Ethnicity: Asian | 1 | 0 | 4 | 0 | 5
  Race/Ethnicity: Hispanic | 42 | 0 | 24 | 0 | 66
  Race/Ethnicity: Non-Hispanic, two or more races | 11 | 0 | 16 | 0 | 27
  Race/Ethnicity: Unknown/Not Reported | 0 | 25 | 0 | 28 | 53
Region of Enrollment [Number; unit: participants]
  United States | 278 | 25 | 232 | 28 | 563
Elementary School Grade [Number; unit: Grade] — Grade in which each student was enrolled Population: Personnel are not included in grade at enrollment as it is not applicable.
  Grade
    Pre-Kindergarten: number analyzed (Participants) | 278 | 0 | 232 | 0 | 510
    Pre-Kindergarten | 19 |  | 0 |  | 19
    Kindergarten: number analyzed (Participants) | 278 | 0 | 232 | 0 | 510
    Kindergarten | 44 |  | 44 |  | 88
    1st Grade: number analyzed (Participants) | 278 | 0 | 232 | 0 | 510
    1st Grade | 40 |  | 39 |  | 79
    2nd Grade: number analyzed (Participants) | 278 | 0 | 232 | 0 | 510
    2nd Grade | 43 |  | 47 |  | 90
    3rd Grade: number analyzed (Participants) | 278 | 0 | 232 | 0 | 510
    3rd Grade | 37 |  | 39 |  | 76
    4th Grade: number analyzed (Participants) | 278 | 0 | 232 | 0 | 510
    4th Grade | 43 |  | 25 |  | 68
    5th Grade: number analyzed (Participants) | 278 | 0 | 232 | 0 | 510
    5th Grade | 52 |  | 38 |  | 90

OUTCOME MEASURES:

1. Primary Outcome: Recruitment of Three 4th or 5th Grade Student Students to Assume the Role as Student Ambassador.
Description: Ability to recruit the required number of 4th or 5th grade student ambassadors at the intervention school at start of trial.
Time Frame: 1 month (pre-intervention to baseline)
Population: Student Ambassadors recruited at the Intervention School, only. Only 3 students were approached for this role and all 3 agreed.
Measure: Count of Participants; unit: Participants
Groups:
- Hydration Intervention - Student Ambassadors: Student ambassadors served as hydration role models, identified "Hydration Heroes", monitored filter lights on hydration stations, & updated the water meter visual throughout the intervention period. They also assisted with the Kick-off event at the start of the intervention.
- Control: Control schools did not have student ambassadors.
Arm/Group | Hydration Intervention - Student Ambassadors | Control
Number analyzed (Participants) | 3 | 0
Participants | 3 | 0

2. Primary Outcome: Retention of 3 Student Ambassadors
Description: Percentage of student ambassadors who continued participation in their role throughout the intervention period (intervention group only).
Time Frame: 4 months
Population: Student ambassadors were recruited in the intervention group only.
Measure: Count of Participants; unit: Participants
Groups:
- Hydration Intervention: Students and staff at the intervention school will receive a school-based hydration intervention that includes a student-developed marketing campaign and incentivizes water bottles in school.
  Hydration Intervention: Teacher & student ambassadors: serve as hydration role models, identify "Hydration Heroes", monitor filter lights on hydration stations, & update the water meter visual.
  Kick-off event: event to kick off the hydration intervention to include water bottles distribution with a station to personalize, experiential activities, and information about the intervention.
  Social marketing: student-developed marketing campaign "Make water your superpower" will be placed in high-traffic areas of the school. Hydration Headquarters will be located in the lunchroom displaying a water meter illustrating bottle refills from the school's hydration stations.
  Behavioral reinforcement: on random days, students drinking water and/or with a water bottle will receive small incentives.
  Education and outreach: Hydration Tip Sheets, hydration signage in classrooms, and hydration trivia on hydration stations. Teachers will deliver 1 hydration lesson per month that align with Standards of Learning.
Arm/Group | Hydration Intervention | Control
Number analyzed (Participants) | 3 | 0
Participants | 3 | 0

3. Primary Outcome: Number of School Personnel Participants Who Reported Being Satisfied With the Intervention
Description: The percent of personnel in the intervention group who agreed or strongly agreed with being satisfied with the intervention (intervention group only). Measured via surveys.
Time Frame: Post (month 4)
Population: Number of staff who completed the survey in the intervention group, only. The number of participants analyzed for this measure is based off the total number of personnel who answered the satisfaction question on the post-intervention [4-month] survey. 25 staff completed some portion of the survey but only 22 answered this specific question.
Measure: Count of Participants; unit: Participants
Groups:
- Hydration Intervention - Staff: Staff at the intervention school will receive a school-based hydration intervention that includes a student-developed marketing campaign and incentivizes water bottles in school.
  Hydration Intervention: Teacher & student ambassadors: serve as hydration role models, identify "Hydration Heroes", monitor filter lights on hydration stations, & update the water meter visual.
  Kick-off event: event to kick off the hydration intervention to include water bottles distribution with a station to personalize, experiential activities, and information about the intervention.
  Social marketing: student-developed marketing campaign "Make water your superpower" will be placed in high-traffic areas of the school. Hydration Headquarters will be located in the lunchroom displaying a water meter illustrating bottle refills from the school's hydration stations.
  Behavioral reinforcement: on random days, students drinking water and/or with a water bottle will receive small incentives.
  Education and outreach: Hydration Tip Sheets, hydration signage in classrooms, and hydration trivia on hydration stations. Teachers will deliver 1 hydration lesson per month that align with Standards of Learning.
  Staff completed a post-intervention survey asked their opinion about the intervention.
- Control: Staff at the control school will participate in assessments only.
Arm/Group | Hydration Intervention - Staff | Control
Number analyzed (Participants) | 22 | 0
Participants | 20 | 0

4. Primary Outcome: Implementation of Intervention Activities.
Description: Percentage of intervention activities conducted per protocol
Time Frame: 4 months
Population: The number of planned core intervention activities that occurred according to protocol (intervention group, only). Activities implemented by teachers, not reported here.
Measure: Count of Units; unit: Core intervention activities
Units Other Than Participants: Core intervention activities
Arm/Group | Hydration Intervention | Control
Number analyzed (Participants) | 303 | 0
Number analyzed (Core intervention activities) | 17 | 0
Core intervention activities | 17 | 0

5. Secondary Outcome: Water Bottle Usage
Description: % of students with water bottles in school
Time Frame: Baseline, mid point 1 (month 2), mid point 2 (month 3), post (month 4)
Population: Number of students enrolled at the school and observed on the assessment date. This number differs from the total student participants at each school due to student absences, therefore were not observed at the observational assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydration Intervention | Control
Number analyzed (Participants) | 240 | 211
Participants
  Baseline: number analyzed (Participants) | 232 | 191
  Baseline | 34 | 17
  Midpoint 1: number analyzed (Participants) | 227 | 211
  Midpoint 1 | 123 | 41
  Midpoint 2 | 113 | 35
  Post: number analyzed (Participants) | 232 | 207
  Post | 120 | 30

6. Secondary Outcome: Hydration Station Usage
Description: Ounces of water used per student per day over 4 months measured by hydration station flow meters. Flow meters captured all water usage in all hydration stations over the 4-month trial. Values were collected from the flow meters at baseline and post (4 months).
Time Frame: Baseline & post (4 month)
Population: Water flowmeters monitored water usage from hydration stations in schools. Hydration station usage is measured by the total amount of ounces of water (across all hydration stations) per student, per school day.
Measure: Number; unit: ounces of water used per student per day
Arm/Group | Hydration Intervention | Control
Number analyzed (Participants) | 278 | 232
ounces of water used per student per day
  Baseline | 0.125 | 0.171
  Post (month 4) | 0.153 | 0.191

7. Secondary Outcome: Sugar-sweetened Beverages at Lunch
Description: % of students with sugar-sweetened beverages at lunch
Time Frame: Baseline, midpoint 1 (month 1), midpoint 2 (month 2), post (month 4)
Population: Number of students enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydration Intervention | Control
Number analyzed (Participants) | 240 | 211
Participants
  Baseline: number analyzed (Participants) | 232 | 191
  Baseline | 33 | 26
  Midpoint 1: number analyzed (Participants) | 227 | 211
  Midpoint 1 | 19 | 30
  Midpoint 2 | 27 | 32
  Post: number analyzed (Participants) | 232 | 207
  Post | 27 | 31

8. Secondary Outcome: Dental Caries Status - Teeth
Description: measured by a modified International Caries Detection and Assessment System (ICDAS) using the DMFT (decayed, missing, and filled permanent teeth)/dmft (decayed, missing, and filled primary teeth) index. DMFT/dmft was defined as the total number of teeth with at least one decayed, missing, or filled tooth surface, with higher scores indicating worse dental health. Possible DMFT (permanent teeth) ranges are 0 to 28. Possible dmft (primary or baby teeth) ranges are 0 to 20.
Time Frame: Baseline and post (month 4)
Population: Number of 3rd grade students who provided assent, with parental consent, to participate in biomedical assessments. If students were not present the day of the assessment, then their data was not captured.
Measure: Median (Full Range); unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Hydration Intervention | Control
Number analyzed (Participants) | 18 | 12
Number analyzed (Teeth) | 12 | 12
Teeth
  Baseline: Decayed Missing and Filled Permanent Teeth: number analyzed (Participants) | 17 | 12
  Baseline: Decayed Missing and Filled Permanent Teeth | 2.0 [0.0 to 6.0] | 2.0 [0.0 to 4.0]
  Baseline: Decayed Missing and Filled Primary Teeth: number analyzed (Participants) | 17 | 12
  Baseline: Decayed Missing and Filled Primary Teeth | 5.0 [0.0 to 12.0] | 1.5 [0.0 to 8.0]
  Post: Decayed Missing and Filled Permanent Teeth: number analyzed (Participants) | 15 | 12
  Post: Decayed Missing and Filled Permanent Teeth | 0.0 [0.0 to 11.0] | 1.5 [0.0 to 5.0]
  Post: Decayed Missing and Filled Primary Teeth: number analyzed (Participants) | 15 | 12
  Post: Decayed Missing and Filled Primary Teeth | 1.0 [0.0 to 12.0] | 3.0 [0.0 to 8.0]

9. Secondary Outcome: Dental Caries Status - Teeth Surfaces
Description: measured by a modified International Caries Detection and Assessment System (ICDAS) using the DMFS (decayed, missing, and filled permanent surfaces)/dmfs (decayed, missing, and filled primary surfaces) index. DMFS/dmfs was defined as the total number of tooth surfaces with decay, fillings, or that were missing due to decay, with higher scores indicating worse dental health. Possible DMFS ranges are 0 to 128 surfaces, as molars and premolars have 5 surfaces and incisors and canines have 4 surfaces, while for baby teeth, possible dmfs ranges from 0-88 surfaces.
Time Frame: Baseline and post (month 4)
Population: as for outcome 8
Measure: Median (Full Range); unit: Teeth Surfaces
Units Other Than Participants: Teeth Surfaces
Arm/Group | Hydration Intervention | Control
Number analyzed (Participants) | 18 | 12
Number analyzed (Teeth Surfaces) | 56 | 56
Teeth Surfaces
  Baseline: Decayed Missing and Filled Surfaces - Permanent Teeth: number analyzed (Participants) | 17 | 12
  Baseline: Decayed Missing and Filled Surfaces - Permanent Teeth: number analyzed (Teeth Surfaces) | 52 | 52
  Baseline: Decayed Missing and Filled Surfaces - Permanent Teeth | 5.0 [0.0 to 14.0] | 3.0 [0.0 to 9.0]
  Baseline: Decayed Missing and Filled Surfaces - Primary Teeth: number analyzed (Participants) | 17 | 12
  Baseline: Decayed Missing and Filled Surfaces - Primary Teeth: number analyzed (Teeth Surfaces) | 56 | 54
  Baseline: Decayed Missing and Filled Surfaces - Primary Teeth | 9.0 [0.0 to 48.0] | 2.0 [0.0 to 40.0]
  Post: Decayed Missing and Filled Surfaces - Permanent Teeth: number analyzed (Participants) | 15 | 12
  Post: Decayed Missing and Filled Surfaces - Permanent Teeth: number analyzed (Teeth Surfaces) | 52 | 52
  Post: Decayed Missing and Filled Surfaces - Permanent Teeth | 1.0 [0.0 to 15.0] | 3.5 [0.0 to 8.0]
  Post: Decayed Missing and Filled Surfaces - Primary Teeth: number analyzed (Participants) | 15 | 12
  Post: Decayed Missing and Filled Surfaces - Primary Teeth: number analyzed (Teeth Surfaces) | 55 | 56
  Post: Decayed Missing and Filled Surfaces - Primary Teeth | 2.0 [0.0 to 46.0] | 5.0 [0.0 to 40.0]

10. Secondary Outcome: Body Mass Index
Description: NHANES Anthropometry methods used to measure height and weight
Time Frame: Baseline and post (month 4)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Hydration Intervention | Control
Number analyzed (Participants) | 18 | 12
kg/m^2
  Baseline | 18.16 (2.90) | 18.7 (2.03)
  Post: number analyzed (Participants) | 15 | 12
  Post | 18.8 (2.86) | 18.70 (2.55)

ADVERSE EVENTS:
Time Frame: Baseline through 4-month assessments (~5 months total).
Groups:
- Hydration Intervention - School Personnel: Staff at the control school will participate in assessments only.
  Control - Assessments Only: Assessments only
Arm/Group | Hydration Intervention - Students | Hydration Intervention - Personnel | Control - Students | Hydration Intervention - School Personnel
All-Cause Mortality (participants affected / at risk) | 0/278 | 0/25 | 0/232 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/278 | 0/25 | 0/232 | 0/28
Other Adverse Events (participants affected / at risk) | 0/278 | 0/25 | 0/232 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-05-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT06132763/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT06132763/SAP_001.pdf